CLINICAL TRIAL: NCT00337753
Title: Cognitive Behavioral Therapy for Pathological Gambling
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Jon E. Grant, University of Minnesota
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0503M68191; K23MH069754-01A1 (NIH)
Record Dates: First submitted 2006-06-14; First posted 2006-06-16 (Estimated); Last update posted 2010-01-05 (Estimated); Status verified 2010-01

CONDITIONS: Pathological Gambling
Keywords: Gambling
MeSH Terms: conditions — Gambling | interventions — Cognitive Behavioral Therapy; Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Behavioral Therapy (Active Comparator): Weekly Cognitive Behavior therapy
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Wait-list (Other): Subjects in wait-list for six-weeks
  Interventions: Behavioral: Wait-list

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — 5-weeks of Cognitive Behavioral Therapy
  Other Names: CBT
  Arms: Cognitive Behavioral Therapy
Behavioral: Wait-list — subjects assigned to wait-list condition for six-weeks
  Arms: Wait-list

SUMMARY:
The purpose of the study is to evaluate a new form of counseling for pathological gambling and to see if the counseling is more effective than attending Gamblers Anonymous.

DETAILED DESCRIPTION:
Subjects will be assigned to counseling or be given a referral list of available Gamblers Anonymous meetings at the first visit based on answers to questions. Assignment to counseling or Gamblers Anonymous will be randomly selected (i.e. chance) with an equal chance of receiving either one. For those assigned to counseling, you will meet with the therapist for 60 minutes weekly. You will receive 5 sessions of counseling.

All subjects will be assessed with gambling questionnaires twice during the 5-week period and again at 3 and 6 months following the 5-week period.

For those assigned to Gamblers Anonymous, they will be offered 5 weeks of counseling at the end of the 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient men and women age 18 to 75
2. Presence of current DSM-IV pathological gambling for at least 6 months duration
3. PG is the most problematic psychiatric disorder (in the patient's and clinician's opinion) and the primary reason for seeking treatment
4. Minimum score of >5 on the South Oaks Gambling Screen which reflects gambling severity consistent with pathological gambling

Exclusion Criteria:

1. Current clinically significant suicidality, severe depression (a score of ≥ 19 on the Hamilton Rating Scale for Depression, 17-item version)(30) or any other disorder requiring immediate intervention
2. Presence of any clinical features requiring a higher level of care than outpatient treatment
3. Cognitive impairment that interferes with the capacity to engage in CBT or to provide informed consent
4. DSM-IV substance abuse or dependence within the past 3 months (see Screening Visit)
5. Current Axis I diagnosis of bipolar disorder or psychotic disorder
6. Previous treatment of CBT for PG (duration of at least 6 sessions); because CBT is not widely used for PG, a minimum of 6 treatments will be rare.
7. Current use of psychotropic medications or within 2 months prior to study entry.
8. Current participation in Gambler's Anonymous (GA).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2006-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
PG-YBOCS | At each visit prior to and after therapy has been completed

SECONDARY OUTCOMES:
Time spent gambling | At each visit prior to and after therapy has been completed

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, MD, JD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States